CLINICAL TRIAL: NCT06700590
Title: (Cost)-Effectiveness of Intensive Trauma-Focused Treatment Versus Spaced Trauma-Focused Treatment As First Line Treatment for Post-Traumatic Stress Disorder in Adults with Multiple Trauma Exposure: Randomized Controlled Trial
Brief Title: First-Line Intervention for PTSD - Intensive Treatment
Acronym: FLIP-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ARQ National Psychotrauma Centre (Other)
Collaborators: Rijksuniversiteit Groningen (Unknown); Psychotraumacentrum Haarlem (Unknown); ARQ IVP BV (Unknown); Militaire GGZ (Unknown); Psy-zo BV (Unknown); Erasmus University Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL86057.018.24; 10390092110006 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-01

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: intensive treatment; massed treatment; randomized controlled trial; RCT; first time treatment
MeSH Terms: conditions — Combat Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: For the clinical interviews (CAPS-5, MINI-S, VLGT), the trained assessors will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- massed/intensive treatment (Experimental)
  Interventions: Behavioral: Intensive Treatment
- spaced/weekly treatment (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Intensive Treatment — Participants engage in two preparatory sessions once weekly, lasting 50 minutes each, which focus on psychoeducation and case conceptualization. The core treatment consists of five days of twice-daily sessions delivered over one or two weeks. The first session of the day consists of prolonged exposure (PE). The second session consists of eye movement desensitization and reprocessing (EMDR). Both treatments are performed in strict adherence to their respective manualized protocol. Two closing sessions focus on lessons learned, integration and a prevention plan. The treatment in total lasts 6 weeks and contains 800 minutes of treatment.
  To enhance practicality, treatment rotation is allowed and encouraged. Rigorous checks on treatment adhenrence will be implemented.
  Arms: massed/intensive treatment
Behavioral: Treatment as usual — Spaced/weekly treatment consists of a treatment-as-usual condition, increasing the representativeness of the control condition. Treatment duration is 800 minutes, either 13 weeks of 60 minutes (with the last sessions being 80 minutes), or 16 weeks of 50 minutes. All evidence-based treatment modalities of the Dutch guidelines are allowed: PE, EMDR, brief eclectic psychotherapy for PTSD (BEPP), narrative exposure therapy (NET), and imaginary rescripting (ImRs). All have common elements of psychoeducation, imaginal exposure, emotional processing, cognitive restructuring and/or meaning making. Treatment adherence will be monitored throughout the intervention. Therapist rotation is not performed
  Arms: spaced/weekly treatment

SUMMARY:
The goal of this clinical trial is to learn if an intensive program can treat post-traumatic stress disorder (PTSD) in adults getting treatment for the first time, and whether it has lower societal costs. The main questions it aims to answer are:

* Does an intensive program reduce PTSD symptoms?
* How expensive is it on a societal level? Researchers will compare the intensive program to the standard weekly treatment to see if the intensive program works to treat PTSD.

Participants will:

* Get 5 days of intensive treatment in two weeks (with two preparatory and closing sessions), or weekly sessions
* Get questionnaires and interviews 5 times in 9 months

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* PTSD diagnosis according to DSM-5 (CAPS-5);
* PTSD diagnosis stemming from 2 or more potentially traumatic events (PTEs)
* seeking first-time treatment for PTSD (or less than 8 sessions);
* employed (working or on sick leave for less than two years)

Exclusion Criteria:

* Current psychotic disorder, severe alcohol or substance use disorder, high suicidal intent (MINI-S for DSM-5) and a concrete suicide plan, or severe aggressive behavior that poses danger for others
* insufficient command of the Dutch language to be able to complete the assessments. This will be determined through clinical judgment at intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  The primary outcome, severity of Post-Traumatic Stress Disorder (PTSD) is assessed by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5). CAPS-5 is a comprehensive 20-item clinical interview that assesses both the DSM-5 PTSD diagnostic criteria and the severity of PTSD symptoms. Scores range from 0 to 80, with higher scores denoting greater symptom severity. The CAPS-5 showed high internal consistency and interrater reliability, good test-retest reliability, and good validity. All the assessors are or will be trained to administer the Dutch versions of the CAPS-5. It requires a total of 225 minutes to complete at all measurement points.
Cost-effectiveness (Quality of life) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Cost-effectiveness is a composite measure of quality of life (physical and mental), and treatment inventory of costs.
  Quality of life will be assessed using the Euro Quality of Life 5 Dimensions (EQ-5D-5L) scale. This scale comprises 14 items categorized into various aspects of health status, rated on a three-point scale.
Cost-effectiveness (Mental Health Quality of Life Questionnaire) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Cost-effectiveness is a composite measure of quality of life (physical and mental), and treatment inventory of costs.
  The Mental Health Quality of Life Questionnaire (MHQoL) will be utilized to assess the quality of life among individuals with mental health issues. The MHQoL comprises a descriptive system (the MHQoL-7D) and a visual analog scale (MHQoL-VAS).
Cost-effectiveness (Treatment inventory of costs) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Cost-effectiveness is a composite measure of quality of life (physical and mental), and treatment inventory of costs. The Treatment Inventory of Costs in Patients with psychiatric disorders (TiC-P) will be utilized to map the costs arising from psychosocial problems in adults. It consists of three components: general questions, questions regarding medical care utilization, and questions related to work.

SECONDARY OUTCOMES:
International Trauma Questionnaire (ITQ) | At baseline (T0).
  The International Trauma Questionnaire (ITQ; Dutch translation) will be used to address the core features of the diagnosis of Post Traumatic Stress Disorder (PTSD) and Complex PTSD (CPTSD) according to the ICD-11 as main study parameter. Several studies have indicated that the preliminary version of the ITQ is a reliable and valid measure of PTSD symptoms. The ITQ assessments will be conducted at all time points, with a total assessment duration of 50 minutes.
Moral Injury Outcome Scale (MIOS) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Moral Injury will be assessed by the Moral Injury Outcome Scale (MIOS). This scale comprises 14 items categorized into two subscales: Shame-Related and Trust-Violation Related Outcomes. It is used to determine if respondents experienced a Potentially Morally Injurious Event (PMIE) and assess the impact of these experiences on well-being. The MIOS also addresses PTSD symptoms related to PMIE. The 14-item MIOS demonstrates invariance and reliability across countries and exhibits two factors: Shame-Related and Trust-Violation-Related Outcomes.
Hospital Anxiety and Depression Scale (HADS) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  The Hospital Anxiety and Depression Scale (HADS) is employed to measure core symptoms of anxiety and depression, excluding physical symptoms. It consists of separate anxiety and depression scales, each with 7 items. The HADS exhibits good homogeneity and test-retest reliability for the total scale and subscales, and its dimensional structure and reliability are stable across different medical settings and age groups.
Acceptance and Action Questionnaire (AAQ-II) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Experiential Avoidance will be assessed by the Experiential Avoidance Assessment (AAQ-II): In its Dutch-language version, the Acceptance and Action Questionnaire-II will be used to assess experiential avoidance. It consists of 7 statements, with higher scores indicating lower experiential avoidance and greater acceptance of unpleasant inner experiences. The Dutch AAQ-II has demonstrated similar construct validity and reliability to the English version.
Personality Inventory for DSM-5-Brief Form-Adult (PID-5-BF-NL) | At baseline (T0), and at 6 months (T3)
  Maladaptive Personality Traits will be assessed by the Personality Inventory for DSM-5-Brief Form-Adult (PID-5-BF-NL). The PID-5-BF-NL will be employed to assess maladaptive personality traits as defined in the alternative DSM-5 model for personality disorders. This self-rated scale comprises 25 items evaluating five personality trait domains. The reliability and validity of the PID-5-BF-NL have demonstrated adequacy to good.
Dissociative Symptoms Assessment (DSS-4) | At baseline (T0), after intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Dissociative Symptoms will be assessed using the Dissociative Symptoms Assessment (DSS-4): The DSS, will be utilized to assess psychoform and somatoform dissociative symptoms experienced in the past week. The scale comprises 21 items and exhibits high internal consistency (Cronbach's alpha = .92) and reliability.
Crisis Support Scale (CSS) | At baseline (T0), after 6 months (T3)
  Social Support will be administered by the Crisis Support Scale (CSS) to evaluate social support, assessing total social support and satisfaction with support. The CSS consists of 7 items and has demonstrated both good validity and reliability. The CSS assessments will be conducted at baseline (T0) and 6 months (T3), with a total assessment duration of 10 minutes.
Verbal Learning and Memory Test (VLGT) | At baseline (T0), after weekly treatment (T2, 17 weeks)
  The Verbal Learning and Memory Test (VLGT), a Dutch version of the American California Verbal Learning Test by Delis, will be employed to assess verbal memory functions in adults. This test evaluates learning performance, speed of learning and forgetting, encoding modes, memorization, recognition over time, sensitivity to interference, the tendency to confabulate, and persistence. The VLGT is a reliable and valid test.
Harms | After intensive treatment (T1, 7 weeks), after weekly treatment (T2, 17 weeks), after 6 months (T3) and 9 months (T4).
  Harms will be assessed by inquiring, 'Have you experienced any issues since your last visit?' following the recommendation by the STRONG STAR consortium.
Treatment satisfaction | at 7 weeks (T1) and 17 weeks (T2)
  Treatment satisfaction will be assessed at 7 weeks (T1) and 17 weeks (T2) for the intensive treatment and treatment as usual, respectively. The Client Satisfaction Questionnaire 8 (CSQ-8) and the Visual Analog Scale will be used. The CSQ-8 is a questionnaire with 8 questions rated on a four-point Likert scale, validated in Dutch samples with high internal consistency and similar psychometric properties to the English version. The Visual Analog Scale with 1 indicating the lowest possible rating and 10 representing the highest possible rating, is utilized for assessing the treatment. Additionally, it includes an inquiry about what modifications or improvements are required to achieve a perfect rating of 10.

OTHER OUTCOMES:
Mini International Neuropsychiatric Interview - Simplified for DSM-5 (MINI-S) | At baseline (T0).
  Diagnoses within the DSM-5 will be assessed using the Mini International Neuropsychiatric Interview - Simplified for DSM-5 (MINI-S; Dutch translation). The MINI-S is a structured diagnostic interview instrument covering the main disorders in DSM-5. The kappa coefficient, sensitivity, and specificity were rated as good to very good for most diagnoses. Inter-rater and test-retest reliability also demonstrated good results.
Life Events Checklist for DSM-5 (LEC-5) | At baseline (T0).
  The Dutch version of The Life Events Checklist for DSM-5 (LEC-5) will be employed at baseline (T0) to assess the types of events experienced by patients for determining trauma exposure in accordance with the DSM-5 to develop the patient case conceptualization. The inventory comprises 57 items where patients respond with either yes or no to indicate their experiences, the age at which the experiences occurred, and their frequency. Although psychometric data for the LEC-5 is not currently available, it is anticipated to exhibit few psychometric differences from the original version, which demonstrates generally adequate psychometric properties.
Adverse Childhood Experience International Questionnaire for adults (ACE-IQ) | At baseline (T0).
  The Adverse Childhood Experience International Questionnaire for adults (ACE-IQ; Dutch translation), a ten-item measure, will be used to assess instances of adverse or traumatic experiences encountered by the patient before reaching the age of 18. The ACE-IQ systematically examines the clients exposure to psychological, physical, and sexual abuse during childhood, as well as household dysfunction. The ACE-IQ demonstrates strong reliability and validity.
Hair cortisol | At baseline (T0).
  Biomarker assessments, i.e. hair cortisol measurement, will be conducted before treatment (T0) with a total assessment duration of 5 minutes. Hair cortisol measurements provide valuable insights into participants' stress levels and physiological responses over time. If the patient objects to sampling the biomarker, this measurement will be dropped, and the patient can participate in the study.
Credibility and Expectancy Questionnaire (CEQ) | At baseline (T0).
  The Credibility and Expectancy Questionnaire (CEQ) will be employed to evaluate patient confidence in the treatment and their perception of the treatment credibility. It employs two response scales and has good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Mink-Nijdam, PhD, Principal Investigator — ARQ National Psychotrauma Center
Locations (4):
- Netherlands (4):
  - ARQ IVP, Diemen, North Holland
  - Psychotraumacentrum Haarlem, Haarlem, North Holland
  - Psy-Zo!, Groningen, Provincie Groningen
  - ARQ Centrum'45, Oegstgeest, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Metadata will be placed in a data repository. IPD can be requested with the research team.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication, at least until 15 years after completion of the trial.
Access Criteria: The IPD can be requested with the first authors by other researchers. Requests will be evaluated on a case-by-case basis. The smallest possible dataset will be delivered, ensuring anonymization of data.

REFERENCES:
- [Derived] Kemmere B, van Pelt YT, Lommen MJJ, Huntjens RJC, Olff M, Mendez MZ, Matthijssen S, Hakkaart-van Roijen L, Nijdam MJ, Heide FJJT. Cost-effectiveness of massed versus spaced trauma-focused treatment as first-line treatment for post-traumatic stress disorder in adults with multiple trauma exposure: protocol for a single-blind non-inferiority randomised controlled trial. BMJ Open. 2025 May 23;15(5):e102530. doi: 10.1136/bmjopen-2025-102530. PMID 40409963